CLINICAL TRIAL: NCT06338384
Title: A Study of Peripheral Neuropathy Clinical Trial Experiences: Insights From Patients
Brief Title: Examining Engagement Trends Among Participants in Peripheral Neuropathy Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 44735129
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Neuropathy
Keywords: peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial aims to uncover the factors driving patient decisions regarding enrollment, withdrawal, or re-engagement in peripheral neuropathy clinical trials. Understanding these factors will significantly improve the relevance and effectiveness of future research endeavors.

Ultimately, this trial endeavors to deepen our understanding of the factors impacting peripheral neuropathy clinical trial participation. Enhancing participation rates could accelerate the development of innovative treatments for this debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Diagnosis of peripheral neuropathy
* Able to comprehend the investigational nature of the protocol and provide informed consent

Exclusion Criteria:

* Female patients who are currently pregnant or nursing
* Inability to perform regular electronic reporting
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral neuropathy who are actively considering enrolling in a clinical study for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of peripheral neuropathy patients who decide to enroll in a clinical research | 3 months
Rate of peripheral neuropathy patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581
- [Background] Lu W, Giobbie-Hurder A, Freedman RA, Shin IH, Lin NU, Partridge AH, Rosenthal DS, Ligibel JA. Acupuncture for Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer Survivors: A Randomized Controlled Pilot Trial. Oncologist. 2020 Apr;25(4):310-318. doi: 10.1634/theoncologist.2019-0489. Epub 2019 Oct 14. PMID 32297442

DOCUMENTS (1):
  • Informed Consent Form (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT06338384/ICF_000.pdf